CLINICAL TRIAL: NCT01474122
Title: Prospective, Randomized, Placebo-controlled, Double-blind, Multicenter, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of Macitentan in Patients With Ischemic Digital Ulcers Associated With Systemic Sclerosis
Brief Title: Macitentan for the Treatment of Digital Ulcers in Systemic Sclerosis Patients
Acronym: DUAL-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: company decision
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC-055C302
Record Dates: First submitted 2011-10-31; First posted 2011-11-18 (Estimated); Results first posted 2015-01-28 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Digital Ulcers
Keywords: digital ulcers; systemic sclerosis
MeSH Terms: conditions — digital ulcers; Scleroderma, Systemic | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Macitentan 3 mg (Active Comparator): Oral macitentan 3 mg, once daily
  Interventions: Drug: Macitentan 3 mg
- Macitentan 10 mg (Active Comparator): Oral macitentan 10 mg, once daily
  Interventions: Drug: Macitentan 10 mg
- Placebo (Placebo Comparator): Oral placebo, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macitentan 3 mg — Macitentan 3-mg tablet once daily
  Other Names: ACT-064992
  Arms: Macitentan 3 mg
Drug: Macitentan 10 mg — Macitentan 10-mg tablet once daily
  Other Names: ACT-064992
  Arms: Macitentan 10 mg
Drug: Placebo — Placebo tablet matching macitentan tablet, once daily
  Arms: Placebo

SUMMARY:
The DUAL-2 study is designed as a multicenter, double-blind two-period study with an initial fixed 16-week Period 1, followed by a Period 2 of variable duration. All patients completing Period 1 continue on their original randomized treatment into Period 2, until the last randomized patient has completed Period 1.

Patients are randomized in a 1:1:1 ratio (macitentan 3mg: macitentan 10mg: placebo).

The primary objective is to demonstrate the effect of macitentan on the reduction of the number of new digital ulcers in patients with systemic sclerosis and ongoing digital ulcers (DU).

Other objectives include:

* the evaluation of the efficacy of macitentan on hand functionality and DU burden at Week 16 in SSc patients with ongoing DU disease.
* the evaluation of the safety and tolerability of macitentan in these patients.
* the evaluation of the efficacy of macitentan on time to first DU complication during the entire treatment period.

DETAILED DESCRIPTION:
Recurrent digital ulcers (DU) are a manifestation of vascular disease in patients with systemic sclerosis (SSc), are an important source of morbidity and lead to impaired function in these patients. In this study, we are investigating whether treatment with the endothelin receptor antagonist, macitentan, decreases the development of new digital ulcers in patients with SSc. Macitentan is a highly potent, tissue-targeting dual endothelin receptor antagonist. Through complete blockade of endothelin action, macitentan is expected to protect tissue from the damaging effect of elevated endothelin. This therapy is not approved for the treatment of systemic sclerosis, but the use of an ERA is an attractive approach in combating the structural vascular damage observed in SSc leading to complications such as DUs.

ELIGIBILITY:
Inclusion Criteria :

* Patients ≥ 18 years of age
* Women of childbearing potential must use two reliable methods of contraception
* Diagnosis of SSc according to the classification criteria of the American College of Rheumatology (ACR)
* At least one visible, active ischemic DU at baseline
* History of at least one additional recent active ischemic digital ulcer

Exclusion Criteria :

* DUs due to condition other than SSc
* Symptomatic pulmonary arterial hypertension (PAH)
* Body mass index (BMI) < 18 kg/m^2
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 x upper limit of normal (ULN)
* Hemoglobin < 75% of the lower limit of the normal range
* Systolic blood pressure < 95 mmHg or diastolic blood pressure < 50 mmHg
* Severe malabsorption; any severe organ failure (e.g., lung, kidney), or any life-threatening condition
* Females who are pregnant or breastfeeding or plan to do so during the course of this study
* Substance or alcohol abuse or dependence, or tobacco use at any level
* Treatment with phosphodiesterase-5 (PDE5) inhibitors
* Patients on statins, who have received treatment for less than 3 months prior to Screening or whose treatment has not been stable during this period
* Patients on vasodilators, who have received treatment for less than 2 weeks prior to Screening or whose treatment has not been stable during this period
* Treatment with prostanoids within 3 months
* Treatment with disease modifying agents if present for less than 3 months prior to Screening or whose treatment has not been stable for at least 1 month prior to Screening
* Treatment with oral corticosteroids (> 10 mg/day of prednisone or equivalent).
* Treatment with endothelin receptor antagonists (ERAs) within 3 months
* Systemic antibiotics to treat infected DU(s) within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

REFERENCES:
- [Result] Khanna D, Denton CP, Merkel PA, Krieg T, Le Brun FO, Marr A, Papadakis K, Pope J, Matucci-Cerinic M, Furst DE; DUAL-1 Investigators; DUAL-2 Investigators. Effect of Macitentan on the Development of New Ischemic Digital Ulcers in Patients With Systemic Sclerosis: DUAL-1 and DUAL-2 Randomized Clinical Trials. JAMA. 2016 May 10;315(18):1975-88. doi: 10.1001/jama.2016.5258. PMID 27163986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 73 centers in 20 countries.The first patient randomized was 9 Feb 2012 and last patient, last visit was 6 Feb 2014.
Pre-assignment Details: A screening visit was performed between Day -14 and Day -1 of the study. Of the 324 patients screened for the study, 59 were screen failures.
Groups:
- Macitentan 3mg: Patients received macitentan once daily at a dose of 3 mg.
- Macitentan 10mg: Patients received macitentan once daily at a dose of 10 mg.
- Placebo: Patients received placebo once daily.
Period: Period 1: Baseline to Week 16
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Started | 88 | 88 (One patient was randomised but did not receive study treatment) | 89
Completed | 87 | 86 | 88
Not Completed | 1 | 2 | 1
Period: Period 2: Week 16 to End of Study
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Started | 87 | 86 | 88
Completed | 70 (Patients on treatment at the time of study termination) | 73 (Patients on treatment at the time of study termination) | 73 (Patients on treatment at the time of study termination)
Not Completed | 17 | 13 | 15

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo | Total
Number analyzed (Participants) | 88 | 88 | 89 | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 76 | 83 | 75 | 234
  >=65 years | 12 | 5 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (13.20) | 47.4 (13.02) | 50.6 (12.88) | 49.6 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 71 | 71 | 217
  Male | 13 | 17 | 18 | 48
Race/Ethnicity, Customized [Number; unit: participants]
  White | 62 | 63 | 68 | 193
  Black or African American | 2 | 0 | 0 | 2
  Asian | 6 | 4 | 6 | 16
  Hispanic | 12 | 14 | 9 | 35
  Other | 6 | 7 | 6 | 19
Region of Enrollment [Number; unit: participants]
  Argentina | 12 | 3 | 3 | 18
  Belgium | 0 | 1 | 0 | 1
  China | 3 | 3 | 5 | 11
  Colombia | 3 | 5 | 6 | 14
  Germany | 2 | 3 | 2 | 7
  Greece | 2 | 4 | 5 | 11
  Ireland | 1 | 2 | 1 | 4
  Israel | 5 | 7 | 12 | 24
  Mexico | 6 | 9 | 6 | 21
  Netherlands | 3 | 2 | 1 | 6
  New Zealand | 2 | 1 | 3 | 6
  Poland | 7 | 11 | 5 | 23
  Portugal | 1 | 2 | 4 | 7
  Puerto Rico | 1 | 1 | 0 | 2
  Russian Federation | 5 | 4 | 7 | 16
  South Africa | 3 | 4 | 2 | 9
  Turkey | 0 | 0 | 1 | 1
  Ukraine | 9 | 7 | 4 | 20
  United Kingdom | 7 | 3 | 6 | 16
  United States | 16 | 16 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of New Digital Ulcers (DUs) up to Week 16
Description: DUs were assessed at each visit starting with the screening visit. Only DUs from the proximal interphalangeal joint (PIP) distally (both on the dorsal and volar surface of the hand, including the digital tip) were recorded. The location of each DU was noted. At each subsequent visit the location of each new DU was noted. DUs that occurred and healed between visits and were reported by patients were not recorded as new DUs. The evaluation was performed by an experienced physician or a trained rater with expertise in the assessment of DUs in systemic sclerosis (SSc). For a given patient, DUs were assessed by the same rater at each visit, whenever possible. Any DU that developed over a previously healed ulcer was recorded as a new DU. Incidence rate is adjusted for 16 weeks of observation, hence is calculated as the number of new DUs/total number of observation days.
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Number; unit: new DUs/16 weeks
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 88 | 88 | 89
new DUs/16 weeks | 1.4413 | 1.3636 | 1.1049
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.434, negative binomial-2 regression (NB-2); NB-2 estimate of new DUs per patient = 1.194, 95% CI 2-sided [0.766 to 1.861] — The estimated value corresponds to the treatment effect i.e. the ratio between the estimated number of new DUs in macitentan 3 mg and in placebo
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.407, NB-2; NB-2 estimate of new DUs per patient = 1.208, 95% CI 2-sided [0.773 to 1.886] — The estimated value corresponds to the treatment effect i.e. the ratio between the estimated number of new DUs in macitentan 10 mg and in placebo

2. Secondary Outcome: Percentage of Participants Without a New DU up to Week 16
Description: DUs were assessed at each visit starting with the screening visit. Only DUs from the proximal interphalangeal joint (PIP) distally (both on the dorsal and volar surface of the hand, including the digital tip) were recorded. The location of each DU was noted. At each subsequent visit the location of each new DU was noted. DUs that occurred and healed between visits and were reported by patients were not recorded as new DUs. The evaluation was performed by an experienced physician or a trained rater with expertise in the assessment of DUs in systemic sclerosis (SSc). For a given patient, DUs were assessed by the same rater at each visit, whenever possible. Any DU that developed over a previously healed ulcer was recorded as a new DU. Numbers of patients with no new DU at Week 16 are imputed using the last observation carried forward method.
Time Frame: Baseline to Week 16
Population: Modified intention to treat set. Ten patients were excluded from the modified intent to treat set due to protocol violations.
Measure: Number; unit: Percentage of participants
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 84 | 84 | 87
Percentage of participants | 56.0 | 54.8 | 59.8
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.5668, Chi-squared; Odds Ratio (OR) = 0.831, 95% CI 2-sided [0.442 to 1.564]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.4624, Chi-squared; Odds Ratio (OR) = 0.789, 95% CI 2-sided [0.420 to 1.484]

3. Secondary Outcome: Percentage of Participants With at Least One DU Complication
Description: DU complications were defined as any one of the following:
  resulting from DU worsening: critical ischemic crisis necessitating hospitalization; gangrene, (auto)amputation; failure of conservative management; surgical and chemical sympathectomy, vascular reconstructions, or any unplanned surgery in the management of hand SSc manifestations; use of parenteral prostanoids; use of endothelin-receptor antagonists; class II, III, or IV narcotics or a > 50% increase in the existing dose compared with baseline; initiation of systemic antibiotics for the treatment of infection attributed to DUs.
Time Frame: Up to 95 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Macitentan 3mg: Patients received macitentan 3mg once daily.
- Macitentan 10mg: Patients received macitentan 10mg once daily.
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 84 | 84 | 87
Percentage of participants | 21.4 | 19.0 | 18.4
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.6117, Chi-squared; Odds Ratio (OR) = 1.216, 95% CI 2-sided [0.572 to 2.582]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.9047, Chi-squared; Odds Ratio (OR) = 1.048, 95% CI 2-sided [0.485 to 2.264]

4. Secondary Outcome: Change in Hand Functionality Health Assessment Questionnaire - Disability Index (HAQ-DI) Hand Component From Baseline to Week 16
Description: HAQ-DI assesses functional ability regarding fine movements of the upper extremities, locomotor activities in the lower extremities, and movements of the upper and lower limbs. Responses were extracted from the Scleroderma Health Assessment Questionnaire covering 8 domains of functional disability (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other daily activities). A mean score ranging from 0-3 was calculated for each domain, and a composite score by dividing the summed domain scores by the number of domains. The composite score was interpreted as 0 (no impairment in function) to 3 (maximal impairment of function). Hand functionality was assessed using a composite of 4 domains (dressing and grooming, grip, hygiene, and eating).
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 84 | 84 | 87
Units on a scale
  Baseline | 1.4 (0.73) | 1.3 (0.70) | 1.4 (0.72)
  Week 16 | 1.2 (0.75) | 1.1 (0.76) | 1.3 (0.77)
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.347, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.165, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.0]

5. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Overall Score From Baseline to Week 16
Description: HAQ-DI assesses functional ability regarding fine movements of the upper extremities, locomotor activities in the lower extremities, and movements of the upper and lower limbs. Responses were extracted from the Scleroderma Health Assessment Questionnaire covering 8 domains of functional disability (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other daily activities). A mean score ranging from 0-3 was calculated for each domain, and a composite score by dividing the summed domain scores by the number of domains. The composite score was interpreted as 0 (no impairment in function) to 3 (maximal impairment of function).
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 84 | 84 | 87
Units on a scale
  Baseline | 1.2 (0.67) | 1.1 (0.65) | 1.2 (0.66)
  Week 16 | 1.1 (0.70) | 1.0 (0.71) | 1.2 (0.68)
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.339, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.312, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

6. Secondary Outcome: Change in Hand Functionality - Hand Disability in Systemic Sclerosis - Digital Ulcers (HDISS-DU) Score From Baseline to Week 16
Description: Patients were asked to answer 24 questions on the use of the hand(s) affected by DUs over the past 7 days on a 6-point scale from 0 (yes without difficulty) to 5 (impossible). The HDISS-DU score is the arithmetic mean of the valid non-missing items. The scores are interpreted as 1 (better ability in completing activities) to 6 (worst ability in completing activities)
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 84 | 84 | 87
Units on a scale
  Baseline | 3.0 (1.08) | 2.9 (1.05) | 2.9 (1.14)
  Week 16 | 2.8 (1.17) | 2.7 (1.11) | 2.9 (1.12)
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.319, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.221, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

ADVERSE EVENTS:
Time Frame: Adverse events occurring during treatment period, up to 95 weeks and up to 30 days after treatment discontinuation
Description: Safety set - all treated patients
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Serious Adverse Events (participants affected / at risk) | 10/88 | 21/87 | 13/89
Other Adverse Events (participants affected / at risk) | 73/88 | 73/87 | 70/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 3mg (N=88) | Macitentan 10mg (N=87) | Placebo (N=89)
INFECTED SKIN ULCER (Infections and infestations) | 1 | 3 | 2
PNEUMONIA (Infections and infestations) | 0 | 2 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 | 1 | 0
GANGRENE (Infections and infestations) | 0 | 1 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
PERITONITIS (Infections and infestations) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 2 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
PARONYCHIA (Infections and infestations) | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
SUBILEUS (Gastrointestinal disorders) | 0 | 1 | 0
ENTERITIS (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 1 | 0
PERICARDITIS (Cardiac disorders) | 0 | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1
DEBRIDEMENT (Surgical and medical procedures) | 0 | 1 | 0
FINGER AMPUTATION (Surgical and medical procedures) | 0 | 1 | 0
IMMUNOSUPPRESSANT DRUG THERAPY (Surgical and medical procedures) | 0 | 1 | 0
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 1 | 0 | 0
SYMPATHECTOMY (Surgical and medical procedures) | 1 | 0 | 1
DRUG THERAPY (Surgical and medical procedures) | 0 | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
SYSTEMIC SCLEROSIS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SCLERODERMA RENAL CRISIS (Renal and urinary disorders) | 0 | 2 | 0
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1 | 1
GLOMERULONEPHRITIS RAPIDLY PROGRESSIVE (Renal and urinary disorders) | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 0
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 | 1 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 | 1 | 0
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 1
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 0
ISCHAEMIC ULCER (General disorders) | 1 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 3mg (N=88) | Macitentan 10mg (N=87) | Placebo (N=89)
HEADACHE (Nervous system disorders) | 17 | 15 | 19
OEDEMA PERIPHERAL (General disorders) | 10 | 14 | 4
DIARRHOEA (Gastrointestinal disorders) | 10 | 10 | 6
NASOPHARYNGITIS (Infections and infestations) | 7 | 10 | 5
ANAEMIA (Blood and lymphatic system disorders) | 6 | 10 | 5
INFECTED SKIN ULCER (Infections and infestations) | 15 | 9 | 13
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 9 | 13
SKIN ULCER (Skin and subcutaneous tissue disorders) | 14 | 8 | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 8 | 6
DIZZINESS (Nervous system disorders) | 5 | 7 | 3
FATIGUE (General disorders) | 2 | 7 | 4
NAUSEA (Gastrointestinal disorders) | 4 | 5 | 2
INFLUENZA (Infections and infestations) | 2 | 5 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 3 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 | 3 | 2
DYSPEPSIA (Gastrointestinal disorders) | 1 | 3 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 2 | 6
CONSTIPATION (Gastrointestinal disorders) | 7 | 2 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 | 2 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6
PHARYNGITIS (Infections and infestations) | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other